CLINICAL TRIAL: NCT02206334
Title: A Phase 1 Study of Stereotactic Body Radiotherapy (SBRT) for the Treatment of Multiple Metastases
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Metastatic Breast Cancer, Non-small Cell Lung Cancer, or Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRG-BR001; NCI-2014-00702 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BR001 (Other: NRG Oncology); NRG-BR001 (Other: CTEP); U10CA180868 (NIH); U10CA021661 (NIH)
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Male Breast Carcinoma; Prostate Adenocarcinoma; Recurrent Breast Carcinoma; Recurrent Non-Small Cell Lung Carcinoma; Recurrent Prostate Carcinoma; Stage IV Breast Cancer; Stage IV Non-Small Cell Lung Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Body Radiation Therapy (SBRT) (Experimental): Patients undergo 3-5 fractions of image-guided stereotactic body radiation therapy to all existing metastases over 1-3 weeks with at least 40 hours between treatments for an individual metastasis.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Undergo SBRT
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; stereotactic radiosurgery; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery; SBRT

SUMMARY:
This phase I trial studies the side effects and the best dose of stereotactic body radiation therapy in treating patients with breast cancer, non-small cell lung cancer, or prostate cancer that has spread to other parts of the body. Stereotactic body radiation therapy delivers fewer, tightly-focused, high doses of radiation therapy to all known sites of cancer in the body while minimizing radiation exposure of surrounding normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended stereotactic body radiation therapy (SBRT) dose for each of the metastatic locations being treated given the individual and overlapping fields when multiple metastases are treated with SBRT in a national clinical trials network setting.

SECONDARY OBJECTIVES:

I. To estimate rates of >= grade 3 Common Terminology Criteria for Adverse Events (CTCAE), version (v.) 4.0 adverse events other than a dose-limiting toxicity (DLT) which is possibly, probably, or definitely related to treatment and which occurs within 6 months from the start of SBRT to multiple metastases.

II. To estimate the rates of long-term adverse events occurring up to 2 years from the end of SBRT.

III. To explore the most appropriate and clinically relevant technological parameters to ensure quality and effectiveness throughout radiation therapy processes, including imaging, simulation, patient immobilization, target and critical structure definition, treatment planning, image guidance and delivery.

OUTLINE:

Patients undergo 3-5 fractions of image-guided stereotactic body radiation therapy to all existing metastases over 1-3 weeks with at least 40 hours between treatments for an individual metastasis.

After completion of study treatment, patients are followed up at 35-45 days and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast cancer (MBC) OR metastatic non-small cell lung cancer (NSCLC) OR metastatic adenocarcinoma of the prostate; the sites of allowed metastases are: peripheral lung, central lung, mediastinal/cervical lymph node, liver, spinal/paraspinal, osseous, and abdominal-pelvic

  * NOTE: after the required number of evaluable patients have been accrued for a given dose level, the accrual for that metastatic location will be temporarily suspended while the safety of that dose level is assessed; a patient can only be entered onto the trial if all of their metastatic locations are open to accrual (e.g. if central lung is temporarily suspended for safety assessment and the patient has a central lung metastases, regardless of other metastases, they cannot enroll until the safety of dose to central lung is determined)
* Primary tumor site without progression at registration
* All metastases not resected must be amenable to SBRT
* The patient must meet ONE of the three following criteria:

  * 3-4 radiographically distinct metastases of any distribution in the allowed anatomical sites OR
  * 2 radiographically distinct metastases that must be anatomically close (i.e., with less than or equal to 5 cm of normal tissue between them) OR
  * 3 or 4 distinct metastasis, 2 or 3 to be treated with SBRT and the other (s) having been surgically removed
* Evaluation by a radiation oncologist within 45 days prior to study registration
* Evaluation by a medical oncologist within 45 days prior to study registration
* The following imaging workup to document metastases within 45 days prior to study registration:

  * Computed tomography (CT) scans of the chest, abdomen and pelvis with radionuclide bone scan OR whole body positron emission tomography (PET)/CT
* History/physical examination within 45 days prior to study registration
* Zubrod performance status =< 2 within 45 days prior to study registration
* Age >= 18 years
* Absolute neutrophil count (ANC) >= 500 cells/mm^3
* Platelets >= 50,000 /mm^3
* Hemoglobin >= 8.0 g/dl (Note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dl is acceptable)
* If liver metastases present, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be < 3 x upper limit of normal (ULN)
* Patient must provide study specific informed consent prior to study entry
* For females of child-bearing potential, negative serum/urine pregnancy test within 14 days prior to study registration

Exclusion Criteria:

* Progression of primary tumor site (breast, prostate, or lung) at time of registration
* Metastases with indistinct borders making targeting not feasible
* Known brain metastases
* Prior palliative radiotherapy to metastases
* Metastases located within 3 cm of the previously irradiated structures:

  * Spinal cord previously irradiated to > 40 Gy (delivered in =< 3 Gy/fraction)
  * Brachial plexus previously irradiated to > 50 Gy (delivered in =< 3 Gy/fraction)
  * Small intestine, large intestine, or stomach previously irradiated to > 45 Gy (delivered in =< 3 Gy/fraction)
  * Brain stem previously irradiated to > 50 Gy (delivered in =< 3 Gy/fraction)
  * Whole lung previously irradiated with prior volume 20 Gy (V20Gy) > 30% (delivered in =< 3 Gy/fraction)
  * Primary tumor irradiated with SBRT
  * Metastasis irradiated with SBRT
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to registration
  * Transmural myocardial infarction within the last 6 months prior to registration
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to registration
  * Severe hepatic disease, defined as a diagnosis of Child-Pugh class B or C hepatic disease
  * Human immunodeficiency virus (HIV) positive with cluster of differentiation (CD) 4 count < 200 cells/microliter; note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count >= 200 cells/microliter within 30 days prior to registration; note also that HIV testing is not required for eligibility for this protocol
  * End-stage renal disease (i.e., on dialysis or dialysis has been recommended)
* Pregnancy or women of childbearing potential not willing/able to use medically acceptable forms of contraception during protocol treatment or for at least 6 months following treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) scored according to the National Cancer Institute (NCI) CTCAE version 4.0 for each of 7 metastatic locations when multiple metastases are treated with SBRT | Within 6 months from the start of treatment; for each of the 7 metastatic locations, analysis occurs after 6 evaluable patients have been followed for a minimum of 6 months from the start of treatment
  Adverse events outlined by metastatic location (full detail in protocol) reported as being probably or definitely related to protocol treatment.

SECONDARY OUTCOMES:
Rate of long-term adverse events, scored according to the NCI CTCAE v. 4.0 | Up to 2 years from end of treatment; analysis occurs after all patients have been potentially followed for 2 years from registration
  Adverse events reported as being possibly, probably, or definitely related to protocol treatment.
Rates of >= grade 3 adverse events, scored according to NCI CTCAE v. 4.0 | Within 6 months from the start of treatment; analysis occurs after all patients have been followed for a minimum of 6 months from the start of treatment
  Adverse events (other than DLTs) reported as being possibly, probably, or definitely related to protocol treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Chmura, Principal Investigator — NRG Oncology
Locations (78):
- United States (73):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Colorado Hospital, Aurora, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Saint Vincent Anderson Regional Hospital/Cancer Center, Anderson, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - GenesisCare USA - Clarkston, Clarkston, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - GenesisCare USA - Farmington Hills, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - GenesisCare USA - Troy, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Virtua Memorial, Mount Holly, New Jersey
  - Cooper CyberKnife Center, Mount Laurel, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Ogden Regional Medical Center, Ogden, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Kantonsspital Aarau, Aarau, Switzerland

REFERENCES:
- [Derived] Chmura S, Winter KA, Robinson C, Pisansky TM, Borges V, Al-Hallaq H, Matuszak M, Park SS, Yi S, Hasan Y, Bazan J, Wong P, Yoon HA, Horton J, Gan G, Milano MT, Sigurdson ER, Moughan J, Salama JK, White J. Evaluation of Safety of Stereotactic Body Radiotherapy for the Treatment of Patients With Multiple Metastases: Findings From the NRG-BR001 Phase 1 Trial. JAMA Oncol. 2021 Jun 1;7(6):845-852. doi: 10.1001/jamaoncol.2021.0687. PMID 33885704